CLINICAL TRIAL: NCT06053346
Title: Evaluation of the Santa Clara County Mental Health Service Pay for Performance Quality Improvement Initiative
Brief Title: Partners in Wellness: Evaluation of a Pay for Performance Program for High-Utilizers of Mental Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Keith Humphreys, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30530
Record Dates: First submitted 2023-08-20; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Psychotic Disorders; Bipolar Disorder; Substance Use Disorders
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Substance-Related Disorders | interventions — Reimbursement, Incentive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pay For Performance (PFP) (Experimental): Participants receive a tailored mix of assertive case management, crisis intervention, substance use counseling, mental health treatment, peer support, skill-building and care coordination, among other services delivered by a provider agency contracted by Santa Clara County. Individual and organizational performance incentives relative to traditional contracted service arrangements were also included. Specifically, the agreement between the contracted provider and the County included an agreed schedule of financial rewards and penalties for the contracted provider based on whether its enrollees utilized more or less care than had a historical cohort of patients enrolled before the program began.
  Interventions: Behavioral: Pay For Performance (PFP)
- Usual Care (UC) (Active Comparator): Participants receive the usual array of mental health and psychosocial services offered by Santa Clara County.
  Interventions: Behavioral: Usual Care (UC)

INTERVENTIONS:
Behavioral: Pay For Performance (PFP) — Wraparound mental health, psychosocial, and addiction treatment services provided by contractor under an schedule of rewards or penalties that was agreed to with Santa Clara County.
  Arms: Pay For Performance (PFP)
Behavioral: Usual Care (UC) — Outpatient and inpatient mental health and psychosocial services delivered by Santa Clara County services and systems.
  Arms: Usual Care (UC)

SUMMARY:
Healthcare systems in the United States (U.S.) have long faced the considerable challenge of managing budgetary pressures while at the same time helping people with serious mental illness and/or addiction. One potential way to address this challenge is to offer community-based services for individuals who are high-utilizers of expensive emergency and inpatient psychiatric services. Due to the decentralized nature of California governance, responsibility for mental health services falls primarily to the individual counties. The County of Santa Clara, CA invests significantly in community-based services as well as 24-hour care settings. This County adopted an innovative Pay for Performance (PFP) model and contracted with a new care provider to better meet the needs of this patient population and, in turn, reduce demand on the County's 24-hour psychiatric services. Whether this innovative contracting framework will help individuals who thus far have not responded well to mental health services is unknown. The purpose of this study was to determine whether the quality of care for these high-need patients was improved and at a sustainable cost. To this end, a randomized clinical trial (RCT) was conducted to determine whether this innovative quality improvement initiative, referred to as "Partners in Wellness", was successful at reducing the total cost of 24-hour psychiatric care used by enrollees compared to individuals who concurrently received services from the county. Individuals were randomly assigned to the Usual Care (UC) or Pay-For-Performance (PFP) conditions. The primary outcome of this evaluation was reduction in the total cost of 24-hour psychiatric services in the target population.

the primary outcome of this evaluation was reduction in the total cost of 24-hour psychiatric services in the target population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a history of extensive utilization of 24-hour psychiatric services in Santa Clara County, CA and a likelihood of continuing to use them in the future.

Exclusion Criteria:

* Age 17 or younger
* Born before 1952
* Not current resident of the County
* Currently residing in a state hospital
* Registered sex offender with legally imposed residency restrictions
* Have a DSM-V diagnosis of (or meet diagnostic criteria for):

  * Dementia
  * Autism Spectrum Disorder
  * Catatonia
  * Brief Psychotic Disorder
  * Traumatic head injury resulting in severe cognitive impairment
  * IQ of 69 or lower
  * Eating disorders, including Pica, Anorexia Nervosa and Bulimia Nervosa, or
  * Pyromania, or Psychogenic Polydipsia paired with life threatening behaviors in the past 12 months.
* Serious risk to self (i.e., suicidal intent with specific plan OR command hallucinations for self-harm that were acted on in the last 30 days and resulted in significant physical injury, or without staff intervention would have resulted in significant physical injury.
* Risk to others (e.g., sexual aggression or other violent, assaultive behavior toward clinical staff in the past 12 months).
* Serious medical diagnoses that either require intensive and regular home health care (e.g., Cystic Fibrosis, Parkinson's, Cancer), imminent risk of placement in a Skilled Nursing Facility or nursing home (e.g., non-ambulatory; needing would care), or are terminal or are life-threatening.
* Significant functional impairments (e.g., unable to toilet, incontinent and refuse to wear diaper, refuse to eat or drink, refuse to dress self or wear clothes, unable to transfer in/out of bed)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Total cost of 24-hour psychiatric services (12 months) | 12 months post-enrollment
  Total cost of the following care types beginning from enrollment until 12 months post-enrollment: Emergency Psychiatric Services (EPS), Barbara Arons Pavilion (BAP) Acute Psychiatric Inpatient, Contract Hospital, Institutes of Mental Disease (IMD), State Hospital, Crisis Residential, Transitional Residential, Super Board and Care, and Residential Care Facility. Days of utilization for each service were multiplied by estimates of the average costs per client, per day provided by the County. To create the primary outcome measure, costs from all of these sources were summed.
Total cost of 24-hour psychiatric services (24 months) | 24 months post-enrollment
  Total cost of the following care types beginning from enrollment until 24 months post-enrollment: Emergency Psychiatric Services (EPS), Barbara Arons Pavilion (BAP) Acute Psychiatric Inpatient, Contract Hospital, Institutes of Mental Disease (IMD), State Hospital, Crisis Residential, Transitional Residential, Super Board and Care, and Residential Care Facility. Days of utilization for each service were multiplied by estimates of the average costs per client, per day provided by the County. To create the primary outcome measure, costs from all of these sources were summed.
Total cost of 24-hour psychiatric services (36 months) | 36 months post-enrollment
  Total cost of the following care types beginning from enrollment until 36 months post-enrollment: Emergency Psychiatric Services (EPS), Barbara Arons Pavilion (BAP) Acute Psychiatric Inpatient, Contract Hospital, Institutes of Mental Disease (IMD), State Hospital, Crisis Residential, Transitional Residential, Super Board and Care, and Residential Care Facility. Days of utilization for each service were multiplied by estimates of the average costs per client, per day provided by the County. To create the primary outcome measure, costs from all of these sources were summed.

SECONDARY OUTCOMES:
Total cost of Barbara Arons Pavilion (BAP) Acute Inpatient Psychiatric Care (12 months) | 12 months post-enrollment
  Total cost of Barbara Arons Pavilion (BAP) Acute Psychiatric Inpatient Care in the 12 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Barbara Arons Pavilion (BAP) Acute Inpatient Psychiatric Care (24 months) | 24 months post-enrollment
  Total cost of Barbara Arons Pavilion (BAP) Acute Psychiatric Inpatient Care in the 24 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Barbara Arons Pavilion (BAP) Acute Inpatient Psychiatric Care (36 months) | 36 months post-enrollment
  Total cost of Barbara Arons Pavilion (BAP) Acute Psychiatric Inpatient Care in the 36 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Emergency Psychiatric Services (EPS) - 12 months | 12 months post-enrollment
  Total cost of Emergency Psychiatric Services (EPS) in the 12 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Emergency Psychiatric Services (EPS) - 24 months | 24 months post-enrollment
  Total cost of Emergency Psychiatric Services (EPS) in the 24 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Emergency Psychiatric Services (EPS) - 36 months | 36 months post-enrollment
  Total cost of Emergency Psychiatric Services (EPS) in the 36 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Contract Hospital (12 months) | 12 months post-enrollment
  Total cost of Contract Hospitals in the 12 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Contract Hospital (24 months) | 24 months post-enrollment
  Total cost of Contract Hospitals in the 24 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Contract Hospital (36 months) | 36 months post-enrollment
  Total cost of Contract Hospitals in the 36 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Crisis Residential Facility (12 months) | 12 months post-enrollment
  Total cost of Crisis Residential Facility care in the 12 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Crisis Residential Facility (24 months) | 24 months post-enrollment
  Total cost of Crisis Residential Facility care in the 24 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Crisis Residential Facility (36 months) | 36 months post-enrollment
  Total cost of Crisis Residential Facility care in the 36 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Transitional Residential (12 months) | 12 months post-enrollment
  Total cost of Transitional Residential care in the 12 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Transitional Residential (24 months) | 24 months post-enrollment
  Total cost of Transitional Residential care in the 24 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Transitional Residential (36 months) | 36 months post-enrollment
  Total cost of Transitional Residential care in the 36 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Residential Care Facility (12 months) | 12 months post-enrollment
  Total cost of Residential Care Facilities in the 12 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Residential Care Facility (24 months) | 24 months post-enrollment
  Total cost of Residential Care Facilities in the 24 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Residential Care Facility (36 months) | 36 months post-enrollment
  Total cost of Residential Care Facilities in the 36 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Institutes of Mental Disease (12 months) | 12 months post-enrollment
  Total cost of Institutes of Mental Disease in the 12 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Institutes of Mental Disease (24 months) | 24 months post-enrollment
  Total cost of Institutes of Mental Disease in the 24 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Institutes of Mental Disease (36 months) | 36 months post-enrollment
  Total cost of Institutes of Mental Disease in the 36 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Custody Health (12 months) | 12 months post-enrollment
  Total cost of Jail-based mental health care in the 12 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Custody Health (24 months) | 24 months post-enrollment
  Total cost of Jail-based mental health care in the 24 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Total cost of Custody Health (36 months) | 36 months post-enrollment
  Total cost of Jail-based mental health care in the 36 months post-enrollment. Days of utilization for this service was multiplied by estimates of the average costs per client, per day provided by the County.
Incarceration (12 months) | 12 months post-enrollment
  Proportion of patients who had any days of incarceration during the 12 months post-enrollment.
Incarceration (24 months) | 24 months post-enrollment
  Proportion of patients who had any days of incarceration during the 24 months post-enrollment.
Incarceration (36 months) | 36 months post-enrollment
  Proportion of patients who had any days of incarceration during the 36 months post-enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Humphreys, PhD, Principal Investigator — Professor of Psychiatry

IPD SHARING:
Plan to Share IPD: No